CLINICAL TRIAL: NCT05171920
Title: A Placebo-Controlled Study of Auxora for the Extended Treatment of High- Risk Patients With Critical COVID-19 Pneumonia (CARDEA-Plus)
Brief Title: A Placebo-Controlled Study of Auxora for the Extended Treatment of High- Risk Patients With Critical COVID-19 Pneumonia
Acronym: CARDEA-Plus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of sufficient numbers of critically ill patients to enroll the study
Sponsor: CalciMedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CM4620-206
Record Dates: First submitted 2021-12-22; First posted 2021-12-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Pneumonia
Keywords: COVID-19; Coronavirus; Pneumonia; Calcium release-activated calcium channel (CRAC) inhibitors; CM4620; Auxora
MeSH Terms: conditions — Pneumonia; COVID-19; Coronavirus Infections | interventions — zegocractin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Auxora (Experimental)
  Interventions: Drug: Auxora
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Auxora — All patients will receive 2.0 mg/kg (1.25 mL/kg) of Auxora at 0 hour and 1.6 mg/kg (1 mL/kg) at both 24 hours and 48 hours from the Start of the First Infusion of Auxora (SFIA) at 0 hour over 4 hours. Patients with severe hypoxemic respiratory failure at 48 hours will be randomized 1:1 to receive extended treatment with Auxora 1.6 mg/kg (1 mL/kg) at 72, 96, and 120 hours from the SFIA
  Arms: Auxora
Drug: Placebo — Patients with severe hypoxemic respiratory failure at 48 hours will be randomized 1:1 to receive 1 mL/kg of Placebo at 72, 96, and 120 hours from the SFIA.
  Arms: Placebo

SUMMARY:
Up to 240 patients with confirmed COVID-19 pneumonia with a baseline imputed PaO2/FiO2 ≤200 receiving oxygen therapy via a high flow nasal cannula (HFNC) or non-invasive ventilation (NIV) will be enrolled at up to 40 sites. All patients will receive three doses of Auxora. Patients who continue to have severe hypoxemic respiratory failure at 48 hours will be randomized to receive three additional doses of Auxora or three doses of placebo. All patients will be followed for 60 days after enrollment into the study.

DETAILED DESCRIPTION:
Up to 240 patients with confirmed COVID-19 pneumonia with a baseline imputed PaO2/FiO2 ≤200 receiving oxygen therapy via a high flow nasal cannula (HFNC) or non-invasive ventilation (NIV) will be enrolled at up to 40 sites. All patients will receive three doses of Auxora.

Patients with severe hypoxemic respiratory failure, those on HFNC with a recorded worst imputed PaO2/FiO2 ≤100 between the end of the infusion of Auxora at 24 hours and the start of the infusion of Auxora at 48 hours or are on NIV or IMV at the start of the infusion of Auxora at 48 hours, will be randomized 1:1 to receive 1.6 mg/kg (1 mL/kg) of Auxora or 1 mL/kg of Placebo at 72, 96 and 120 hours from the SFIA. Patients on IMV will be stratified between the Auxora and Placebo groups. Patients without severe hypoxemic respiratory failure, those with a recorded worst imputed PaO2/FiO2 >100 between the end of the infusion of Auxora at 24 hours and the start of the infusion of Auxora at 48 hours and are not on NIV or IMV, will not be randomized for further infusions but will remain in the study and complete all assessments through Day 60.

Patients enrolled in the study should receive dexamethasone, or equivalent dose of another corticosteroid, as standard of care. The use of remdesivir should be considered and the use of tocilizumab is encouraged.

ELIGIBILITY:
Inclusion Criteria:

1. Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay in any specimen, as documented by either of the following:

   * PCR positive in sample collected < 72 hours prior to consent;
   * PCR positive in sample collected ≥ 72 hours prior to consent, with inability to obtain a repeat sample (e.g. due to lack of testing supplies, or limited testing capacity, or results taking >24 hours, etc.) or progressive disease suggestive of ongoing SARS-CoV-2 infection;
2. At least 1 of the following symptoms:

   o Fever, cough, sore throat, malaise, headache, muscle pain, dyspnea at rest or with exertion, confusion, or respiratory distress;
3. A PaO2/FiO2 ≤200 recorded in the 24 hours before consent. The PaO2/FiO2 can be imputed from pulse oximetry;
4. Oxygen therapy being administered via HFNC or NIV
5. The presence of a respiratory infiltrate or abnormality consistent with pneumonia that is documented by either a CXR or CT scan of the lungs;
6. The patient is ≥18 years of age;
7. A female patient of childbearing potential must not attempt to become pregnant for 180 days, and if sexually active with a male partner, is willing to practice acceptable methods of birth control for 180 days after the last dose of study drug;
8. A male patient who is sexually active with a female partner of childbearing potential is willing to practice acceptable methods of birth control for 180 days after the last dose of study drug. A male patient must not donate sperm for 180 days;
9. The patient is willing and able to, or has a legal authorized representative (LAR) who is willing and able to, provide informed consent to participate, and to cooperate with all aspects of the protocol.

Exclusion Criteria:

1. Do Not Intubate order;
2. PaO2/FiO2 ≤75 recorded at the time of consent. The PaO2/FiO2 can be imputed from pulse oximetry;
3. Receiving IMV via endotracheal intubation or tracheostomy;
4. Receiving ECMO;
5. Shock defined by the use of vasopressors;
6. Known history of:

   * Organ or hematologic transplant;
   * HIV;
   * Active hepatitis B, or hepatitis C infection;
7. Current treatment with:

   * Chemotherapy;
   * Immunosuppressive medications or immunotherapy (see protocol (Section 5.3) for list of prohibited immunosuppressive medications and immunotherapy) at the time of consent;
   * Hemodialysis or Peritoneal Dialysis;
8. Known to be pregnant or is nursing;
9. Currently participating in another study of an investigational drug or therapeutic medical device at the time of consent;
10. Known allergy to eggs or any of the excipients in study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of randomized patients receiving 6 versus 3 doses of Auxora requiring IMV or dying after 72 hours from the SFIA through day 60. | SFIA through day 60

SECONDARY OUTCOMES:
All-Cause Mortality in randomized patients receiving 6 versus 3 doses of Auxora | SFIA through day 60
All-Cause Mortality in randomized patients receiving 6 versus 3 doses of Auxora | SFIA through day 30
Proportion of randomized patients receiving 6 versus 3 doses of Auxora requiring IMV after 72 hours | SFIA through day 60
Number of Days in the Hospital | Hospital admission through discharge from hospital
Number of Days in the ICU | Hospital admission through discharge from the ICU
The incidence of TEAEs and SAEs | From SFIA through day 60
The intensity and relationship of TEAEs and SAEs | From SFIA through day 60

OTHER OUTCOMES:
Exploratory: Difference in Angiopoietin 2 levels after treatment with Auxora | Baseline through 192 hours
Exploratory: Difference in Angiopoietin 1 level after treatment with Auxora | Baseline through 192 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Hebbar, MD, Study Director — CalciMedica, Inc.
Locations (3):
- United States (3):
  - Regions Hospital, Saint Paul, Minnesota
  - Methodist Hospital, Saint Paul, Minnesota
  - JPS Health, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No